CLINICAL TRIAL: NCT01208207
Title: A Phase III, Two-Part, Randomized, Double-Blind, Active Comparator-Controlled, Multicenter Clinical Trial to Study the Relative Efficacy and Tolerability of Two Doses of MK-0663/Etoricoxib in Patients With Ankylosing Spondylitis
Brief Title: A Two-Part 26-Week Study of Etoricoxib as Treatment for Ankylosing Spondylitis (AS) (MK-0663-108)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0663-108
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- etoricoxib 60 mg/etoricoxib 60 mg (Experimental): The etoricoxib 60 mg/etoricoxib 60 mg treatment sequence will receive etoricoxib 60 mg in Part I and Part II
  Interventions: Drug: Part I - etoricoxib 60 mg; Drug: Part I - Placebo to naproxen 500 mg; Drug: Part II- etoricoxib 60 mg; Drug: Part I - Placebo to etoricoxib 90 mg; Drug: Part II - Placebo to etoricoxib 90 mg; Drug: Part II- Placebo to naproxen 500 mg
- etoricoxib 60 mg/etoricoxib 90 mg (Experimental): The etoricoxib 60 mg/etoricoxib 90 mg treatment sequence will receive etoricoxib 60 mg in Part I and etoricoxib 90 mg in Part II
  Interventions: Drug: Part I - etoricoxib 60 mg; Drug: Part I - Placebo to naproxen 500 mg; Drug: Part II- etoricoxib 90 mg; Drug: Part I - Placebo to etoricoxib 90 mg; Drug: Part II- Placebo to etoricoxib 60 mg; Drug: Part II- Placebo to naproxen 500 mg
- etoricoxib 90 mg/etoricoxib 90 mg (Experimental): The etoricoxib 90 mg/etoricoxib 90 mg treatment sequence will receive etoricoxib 90 mg in Part I and Part II
  Interventions: Drug: Part I - etoricoxib 90 mg; Drug: Part I - Placebo to naproxen 500 mg; Drug: Part II- etoricoxib 90 mg; Drug: Part I - Placebo to etoricoxib 60 mg; Drug: Part II- Placebo to etoricoxib 60 mg; Drug: Part II- Placebo to naproxen 500 mg
- naproxen 1000 mg/naproxen 1000 mg (Active Comparator): The naproxen 1000 mg/naproxen 1000 mg treatment sequence will receive naproxen 1000 mg in Part I and Part II
  Interventions: Drug: Part I- naproxen 1000 mg; Drug: Part II- naproxen 1000 mg; Drug: Part I - Placebo to etoricoxib 60 mg; Drug: Part I - Placebo to etoricoxib 90 mg; Drug: Part II- Placebo to etoricoxib 60 mg; Drug: Part II - Placebo to etoricoxib 90 mg

INTERVENTIONS:
Drug: Part I - etoricoxib 60 mg — etoricoxib 60 mg oral tablet once daily for 6 weeks
  Other Names: MK-0663
  Arms: etoricoxib 60 mg/etoricoxib 60 mg; etoricoxib 60 mg/etoricoxib 90 mg
Drug: Part I - etoricoxib 90 mg — etoricoxib 90 mg oral tablet once daily for 6 weeks
  Other Names: Mk-0663
  Arms: etoricoxib 90 mg/etoricoxib 90 mg
Drug: Part I- naproxen 1000 mg — naproxen 500 mg oral tablet twice daily for 6 weeks
  Arms: naproxen 1000 mg/naproxen 1000 mg
Drug: Part I - Placebo to naproxen 500 mg — Placebo to naproxen 500 mg oral tablet twice daily for 6 weeks
  Arms: etoricoxib 60 mg/etoricoxib 60 mg; etoricoxib 60 mg/etoricoxib 90 mg; etoricoxib 90 mg/etoricoxib 90 mg
Drug: Part II- etoricoxib 60 mg — etoricoxib 60 mg oral tablet once daily for 20 weeks
  Other Names: MK-0663
  Arms: etoricoxib 60 mg/etoricoxib 60 mg
Drug: Part II- etoricoxib 90 mg — etoricoxib 90 mg oral tablet once daily for 20 weeks
  Other Names: MK-0663
  Arms: etoricoxib 60 mg/etoricoxib 90 mg; etoricoxib 90 mg/etoricoxib 90 mg
Drug: Part II- naproxen 1000 mg — naproxen 500 mg oral tablet twice daily for 20 weeks
  Arms: naproxen 1000 mg/naproxen 1000 mg
Drug: Part I - Placebo to etoricoxib 60 mg — Placebo to etoricoxib 60 mg oral tablet once daily for 6 weeks.
  Arms: etoricoxib 90 mg/etoricoxib 90 mg; naproxen 1000 mg/naproxen 1000 mg
Drug: Part I - Placebo to etoricoxib 90 mg — Placebo to etoricoxib 90 mg oral tablet once daily for 6 weeks.
  Arms: etoricoxib 60 mg/etoricoxib 60 mg; etoricoxib 60 mg/etoricoxib 90 mg; naproxen 1000 mg/naproxen 1000 mg
Drug: Part II- Placebo to etoricoxib 60 mg — Placebo to etoricoxib 60 mg oral tablet once daily for 20 weeks.
  Arms: etoricoxib 60 mg/etoricoxib 90 mg; etoricoxib 90 mg/etoricoxib 90 mg; naproxen 1000 mg/naproxen 1000 mg
Drug: Part II - Placebo to etoricoxib 90 mg — Placebo to etoricoxib 90 mg oral tablet once daily for 20 weeks.
  Arms: etoricoxib 60 mg/etoricoxib 60 mg; naproxen 1000 mg/naproxen 1000 mg
Drug: Part II- Placebo to naproxen 500 mg — Placebo to naproxen 500 mg orally twice daily for 20 weeks.
  Arms: etoricoxib 60 mg/etoricoxib 60 mg; etoricoxib 60 mg/etoricoxib 90 mg; etoricoxib 90 mg/etoricoxib 90 mg

SUMMARY:
The purpose of the study is to evaluate the efficacy and tolerability of two doses of etoricoxib compared to naproxen in the treatment of ankylosing spondylitis (AS). The primary objectives are to evaluate the improvement in Spinal Pain Intensity over 6 weeks of treatment with etoricoxib 90 mg or 60 mg compared to naproxen; and to evaluate the improvement in Spinal Pain Intensity over 6 weeks of treatment with etoricoxib 90 mg compared with etoricoxib 60 mg. Additionally the added benefit of increasing the dose of etoricoxib from 60 mg to 90 mg will be assessed in the second part of the study. The primary hypothesis is that the improvement in Spinal Pain Intensity visual analog scale (VAS) as measured by the time-weighted average (TWA) change from baseline over 6 weeks of treatment in Part I for etoricoxib 90 mg or 60 mg once daily is not inferior to naproxen 1000 mg.

ELIGIBILITY:
Inclusion Criteria:

* Has a definite diagnosis of Ankylosing Spondylitis (AS) per Modified New York Criteria made at least 6 months prior to screening
* Has a history of positive therapeutic benefit with non-steroidal anti-inflammatory drugs (NSAIDs) and regular use of NSAIDS for past 30 days
* Has a score on Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Question 2 at screening visit that is <77 mm
* Must demonstrate sufficient "flare" or worsening of AS pain
* Is in general good health (other than AS)
* Has had approved non-study antirheumatic therapy that has been at stable dosing AND is not anticipated to undergo a change within the first 6 weeks of the protocol

Exclusion Criteria:

* Has inflammatory arthritis (eg, rheumatoid arthritis, psoriatic arthritis, crystal-induced arthritis, spondyloarthropathy, diffuse idiopathic skeletal hyperostosis [DISH]), polymyalgia rheumatica, a history of septic arthritis or intra-articular fracture of the study joint, Wilson's disease, hemachromatosis, ochronosis, or primary osteochondromatosis
* Has acute peripheral articular disease (onset within 4 weeks prior to screening) of an active (painful or swollen) peripheral arthritis
* Has a history of gastric or biliary surgery, or small intestine surgery that causes clinical malabsorption
* Has had an active peptic (gastric or duodenal) ulcer or history of inflammatory bowel disease
* Has undergone coronary artery bypass graft surgery (CABG), angioplasty, or has a cerebrovascular accident or transient ischemic attack within the past 6 months or has active ischemic heart disease, cerebrovascular disease, or peripheral vascular disease
* Has Class II-IV congestive heart failure
* Has uncontrolled hypertension
* Has a history of neoplastic disease, except adequately treated basal cell carcinoma or carcinoma in situ of the cervix, or malignancies that have been successfully treated ≥ 5 years prior to screening
* Has history of leukemia, lymphoma, malignant melanoma, and myeloproliferative disease
* Allergy to etoricoxib or naproxen, or history of a significant clinical or laboratory adverse experience associated with etoricoxib or naproxen
* Has a history or family history of an inherited or acquired bleeding disorder
* Is considered morbidly obese and demonstrates significant health problems stemming from obesity, which would confound study participation or interpretation of study results
* Is pregnant, breast-feeding, or expecting to conceive during the study
* Has a clinical diagnosis of hepatic insufficiency defined as Child-Pugh score ≥ 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2010-09-27 (Actual); Primary Completion 2014-11-12 (Actual); Study Completion 2014-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Balazcs E, Sieper J, Bickham K, Mehta A, Frontera N, Stryszak P, Popmihajlov Z, Peloso PM. A randomized, clinical trial to assess the relative efficacy and tolerability of two doses of etoricoxib versus naproxen in patients with ankylosing spondylitis. BMC Musculoskelet Disord. 2016 Oct 13;17(1):426. doi: 10.1186/s12891-016-1275-5. PMID 27737664

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All Patients Randomized
Groups:
- Etoricoxib 60 mg (Part I): Etoricoxib 60 mg oral tablet once daily for 6 weeks
- Etoricoxib 90 mg (Part I): Etoricoxib 90 mg oral tablet once daily for 6 weeks
- Naproxen 1000 mg (Part I): Naproxen 500 mg oral tablet twice daily for 6 weeks
- Etoricoxib 60 mg / 60 mg (Part II): A continuation of the etoricoxib 60 mg oral tablet once daily for 20 weeks (Part II)
- Etoricoxib 60 mg / 90 mg (Part II): An increase of etoricoxib to 90 mg for 20 weeks (Part II)
- Etoricoxib 90 mg / 90 mg (Part II): A continuation of the etoricoxib 90 mg oral tablet once daily for 20 weeks (Part II)
- Naproxen 1000 mg (Part II): A continuation of the naproxen 500 mg oral tablet twice daily for 20 weeks (Part II)
Period: Part I
Arm/Group | Etoricoxib 60 mg (Part I) | Etoricoxib 90 mg (Part I) | Naproxen 1000 mg (Part I) | Etoricoxib 60 mg / 60 mg (Part II) | Etoricoxib 60 mg / 90 mg (Part II) | Etoricoxib 90 mg / 90 mg (Part II) | Naproxen 1000 mg (Part II)
Started | 702 | 156 | 157 | 0 | 0 | 0 | 0
Completed | 632 | 145 | 142 | 0 | 0 | 0 | 0
Not Completed | 70 | 11 | 15 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 19 | 2 | 6 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 21 | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance With Study Drug | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 8 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 14 | 4 | 4 | 0 | 0 | 0 | 0
Period: Part II
Arm/Group | Etoricoxib 60 mg (Part I) | Etoricoxib 90 mg (Part I) | Naproxen 1000 mg (Part I) | Etoricoxib 60 mg / 60 mg (Part II) | Etoricoxib 60 mg / 90 mg (Part II) | Etoricoxib 90 mg / 90 mg (Part II) | Naproxen 1000 mg (Part II)
Started | 0 | 0 | 0 | 314 | 318 | 145 | 142
Completed | 0 | 0 | 0 | 282 | 295 | 129 | 131
Not Completed | 0 | 0 | 0 | 32 | 23 | 16 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 10 | 9 | 3 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 5 | 9 | 4 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 6 | 4 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4 | 0 | 2 | 1
Not completed — Non-Compliance With Study Drug | 0 | 0 | 0 | 4 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Technical Problems | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Etoricoxib 60 mg: Etoricoxib 60 mg oral tablet once daily
- Etoricoxib 90 mg: Etoricoxib 90 mg once daily
- Naproxen 1000 mg: Naproxen 500 mg oral tablet twice daily
- Total: Total of all reporting groups
Arm/Group | Etoricoxib 60 mg | Etoricoxib 90 mg | Naproxen 1000 mg | Total
Number analyzed (Participants) | 702 | 156 | 157 | 1015
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.4 (12.4) | 45.2 (11.3) | 44.5 (12.3) | 45.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 45 | 41 | 295
  Male | 493 | 111 | 116 | 720
Spinal Pain Intensity [Mean (Standard Deviation); unit: mm VAS] — Visual Analogue Scale from 0-100 mm with a lower value representing a better response.
  mm VAS | 76.7 (14.2) | 76.7 (15.2) | 77.0 (14.0) | 76.8 (14.3)

OUTCOME MEASURES:

1. Primary Outcome: Time-Weighted Average Change From Baseline in the Spinal Pain Intensity in Study Part 1: Etoricoxib 90 mg vs. Naproxen
Description: Spinal Pain Intensity is measured using a visual analog scale (VAS) from 0-100 mm with a lower value representing a better response. The time-weighted average change is calculated by taking the time between adjacent observations divided by the time from the randomization visit to the last observation in the period of interest, and using it as the weight for computation of the average.
Time Frame: Baseline and up to Week 6
Population: Per-Protocol Population - excluded participants due to important protocol deviations that may have had a substantial effect on the result of the primary efficacy endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm VAS
Groups:
- Etoricoxib 90 mg: Etoricoxib 90 mg oral tablet once daily for 6 weeks
- Naproxen 1000 mg: Naproxen 500 mg oral tablet twice daily for 6 weeks
Arm/Group | Etoricoxib 90 mg | Naproxen 1000 mg
Number analyzed (Participants) | 144 | 143
mm VAS | -31.23 [-34.70 to -27.76] | -30.59 [-34.07 to -27.10]
Statistical Analysis 1: Comparison: Etoricoxib 90 mg vs Naproxen 1000 mg; Test type: Non-Inferiority or Equivalence — The etoricoxib dose (90 mg) will be considered non-inferior to naproxen 1000 mg if the upper bound of the two-sided 95% confidence interval of the between-treatment difference in the least squares (LS) mean (etoricoxib minus naproxen 1000 mg) is no larger than 8 mm VAS (non-inferiority margin); ANCOVA; Difference in Least Squares Mean = -0.64, 95% CI 2-sided [-5.47 to 4.19]

2. Primary Outcome: Time-Weighted Average Change From Baseline in the Spinal Pain Intensity in Study Part 1: Etoricoxib 60 mg vs. Naproxen
Description: as for outcome 1
Time Frame: Baseline and up to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm VAS
Groups:
- Etoricoxib 60 mg: Etoricoxib 60 mg oral tablet once daily for 6 weeks
Arm/Group | Etoricoxib 60 mg | Naproxen 1000 mg
Number analyzed (Participants) | 660 | 143
mm VAS | -29.00 [-30.69 to -27.31] | -30.59 [-34.07 to -27.10]
Statistical Analysis 1: Comparison: Etoricoxib 60 mg vs Naproxen 1000 mg; Test type: Non-Inferiority or Equivalence — The etoricoxib dose (60 mg) will be considered non-inferior to naproxen 1000 mg if the upper bound of the two-sided 95% confidence interval of the between-treatment difference in the LS mean (etoricoxib minus naproxen 1000 mg) is no larger than 8 mm VAS (non-inferiority margin); ANCOVA; Difference in Least Squares Mean = 1.59, 95% CI 2-sided [-2.19 to 5.37]

3. Secondary Outcome: Time-Weighted Average Change From Baseline in the Spinal Pain Intensity in Study Part 1: Etoricoxib 90 mg vs. Etoricoxib 60 mg
Description: as for outcome 1
Time Frame: Baseline and up to Week 6
Population: Modified Intent-to-Treat (mITT) Population - the mITT population in Part I consisted of all randomized participants who received at least 1 dose of study treatment, had at least 1 measurement of interest post-randomization that was collected within 3 days of the last dose of study medication taken in Part I, and had baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm VAS
Arm/Group | Etoricoxib 90 mg | Etoricoxib 60 mg
Number analyzed (Participants) | 153 | 694
mm VAS | -30.51 [-33.87 to -27.15] | -28.94 [-30.58 to -27.29]
Statistical Analysis 1: Comparison: Etoricoxib 90 mg vs Etoricoxib 60 mg; Test type: Superiority or Other; p = 0.396, ANCOVA; Difference in Least Squares Mean = -1.58, 80% CI 2-sided [-3.96 to 0.81]

4. Secondary Outcome: Average Change From Week 6 in the Spinal Pain Intensity Over Weeks 10 and 12 in Study Part 2: Etoricoxib 60/90 mg vs. Etoricoxib 60mg (Non-responders From Part I)
Description: Spinal Pain Intensity is measured using a visual analog scale (VAS) from 0-100 mm with a lower value representing a better response. Average change from Week 6 in Spinal Pain Intensity (VAS) over Weeks 10 and 12 is calculated as the average Spinal pain Intensity (VAS) value over Weeks 10 and 12 minus the Spinal Pain Intensity (VAS) at Week 6.
Time Frame: Week 6 to Week 10 and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: mm VAS
Groups:
- Etoricoxib 60 mg/ 90 mg: Etoricoxib 60 mg in Part I and Etoricoxib 90 mg in Part II
- Etoricoxib 60 mg / 60 mg: Etoricoxib 60 mg in Part I and Etoricoxib 60 mg in Part II
Arm/Group | Etoricoxib 60 mg/ 90 mg | Etoricoxib 60 mg / 60 mg
Number analyzed (Participants) | 178 | 175
mm VAS | -9.97 [-12.42 to -7.51] | -7.26 [-9.73 to -4.80]
Statistical Analysis 1: Comparison: Etoricoxib 60 mg/ 90 mg vs Etoricoxib 60 mg / 60 mg; Test type: Superiority or Other; p = 0.112, ANCOVA; Difference in Least Squares Mean = -2.70, 80% CI [-4.88 to -0.52]

5. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to an Adverse Event
Time Frame: Up to 26 weeks
Population: All Patients as Treated Population (APaT) - Participants were included in the treatment group corresponding to the study treatment they actually received. One participant randomized to 60 mg in Part II received 90 mg in Part II, and; therefore, was included in the Etoricoxib 60mg / 90mg (Part II) arm.
Measure: Number; unit: Participants
Arm/Group | Etoricoxib 60 mg (Part I) | Etoricoxib 90 mg (Part I) | Naproxen 1000 mg (Part I) | Etoricoxib 60 mg / 60 mg (Part II) | Etoricoxib 60 mg / 90 mg (Part II) | Etoricoxib 90 mg / 90 mg (Part II) | Naproxen 1000 mg (Part II)
Number analyzed (Participants) | 702 | 155 | 156 | 313 | 319 | 145 | 142
Participants | 22 | 2 | 6 | 3 | 9 | 4 | 2

ADVERSE EVENTS:
Time Frame: Up to Week 30 (including up to 28 days after last dose of study drug)
Description: AE's were collected for the All Patients as Treated Population. Participants were included in the treatment group corresponding to the study treatment they actually received. One participant randomized to Etoricoxib 60 mg in Part II received Etoricoxib 90 mg in Part II, and; therefore, was included in the Etoricoxib 60mg / 90mg (Part II) arm.
Groups:
- Etoricoxib 60 mg / Etoricoxib 60 mg: Participants who received Etoricoxib 60 mg in Part I and at least one dose of Etoricoxib 60 mg in Part II.
- Etoricoxib 60 mg / Etoricoxib 90 mg: Participants who received Etoricoxib 60 mg in Part I and at least one dose of Etoricoxib 90 mg in Part II.
- Etoricoxib 90 mg / Etoricoxib 90 mg: Participants who received Etoricoxib 90 mg in Part I and at least one dose of Etoricoxib 90 mg in Part II.
- Naproxen 1000 mg / Naproxen 1000 mg: Participants who received Naproxen 1000 mg in Part I and at least one dose of Naproxen 1000 mg in Part II.
- Etoricoxib 60 mg: Participants who received at least one dose of Etoricoxib 60 mg in Part I, but no drug in Part II.
- Etoricoxib 90 mg: Participants who received at least one dose of Etoricoxib 90 mg in Part I, but no drug in Part II.
- Naproxen 1000 mg: Participants who received at least one dose of Naproxen 1000 mg in Part I, but no drug in Part II.
Arm/Group | Etoricoxib 60 mg / Etoricoxib 60 mg | Etoricoxib 60 mg / Etoricoxib 90 mg | Etoricoxib 90 mg / Etoricoxib 90 mg | Naproxen 1000 mg / Naproxen 1000 mg | Etoricoxib 60 mg | Etoricoxib 90 mg | Naproxen 1000 mg
Serious Adverse Events (participants affected / at risk) | 1/313 | 7/319 | 6/145 | 2/142 | 5/70 | 0/10 | 0/14
Other Adverse Events (participants affected / at risk) | 55/313 | 50/319 | 24/145 | 25/142 | 18/70 | 6/10 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib 60 mg / Etoricoxib 60 mg (N=313) | Etoricoxib 60 mg / Etoricoxib 90 mg (N=319) | Etoricoxib 90 mg / Etoricoxib 90 mg (N=145) | Naproxen 1000 mg / Naproxen 1000 mg (N=142) | Etoricoxib 60 mg (N=70) | Etoricoxib 90 mg (N=10) | Naproxen 1000 mg (N=14)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib 60 mg / Etoricoxib 60 mg (N=313) | Etoricoxib 60 mg / Etoricoxib 90 mg (N=319) | Etoricoxib 90 mg / Etoricoxib 90 mg (N=145) | Naproxen 1000 mg / Naproxen 1000 mg (N=142) | Etoricoxib 60 mg (N=70) | Etoricoxib 90 mg (N=10) | Naproxen 1000 mg (N=14)
Abdominal pain upper (Gastrointestinal disorders) | 15 (28) | 8 (12) | 2 (2) | 10 (10) | 3 (6) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 17 (19) | 21 (21) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 10 (15) | 13 (18) | 9 (11) | 5 (5) | 4 (13) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 18 (21) | 15 (16) | 8 (8) | 8 (8) | 4 (4) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 7 (8) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 8 (8) | 2 (2) | 4 (5) | 4 (6) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (4) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 9 (10) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 4 (10) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.